CLINICAL TRIAL: NCT03192033
Title: STEP: Proglide® Versus Femoseal®: A Randomized Controlled Trial to Compare the Efficacy of Arterial Closure Devices Following Endovascular Peripheral Arterial Procedures
Brief Title: STEP: Proglide® Versus Femoseal®: A Trial to Compare the Efficacy of Arterial Closure Devices Following Endovascular Peripheral Arterial Procedures
Acronym: STEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC16_0466
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Intervention Model Description: A duplex scan guided retrograde femoral puncture is performed followed by the use of a closure arterial device to ensure hemostasis. Patients are randomly assigned to be closed by Proglide® (Abbott) versus Femoseal® (Terumo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arterial closure device used is Proglide® (Abbott) (Other)
  Interventions: Other: Arterial closure to ensure hemostasis at femoral artery puncture points; Device: Proglide® (Abbott)
- Arterial closure device used is Femoseal® (Terumo) (Other)
  Interventions: Device: Femoseal® (Terumo); Other: Arterial closure to ensure hemostasis at femoral artery puncture points

INTERVENTIONS:
Other: Arterial closure to ensure hemostasis at femoral artery puncture points — Arterial closure devices used: Proglide® (Abbott)
  Arms: Arterial closure device used is Proglide® (Abbott)
Device: Proglide® (Abbott) — Arterial closure device used: Proglide® (Abbott)
  Arms: Arterial closure device used is Proglide® (Abbott)
Device: Femoseal® (Terumo) — Arterial closure device used: Femoseal® (Terumo)
  Arms: Arterial closure device used is Femoseal® (Terumo)
Other: Arterial closure to ensure hemostasis at femoral artery puncture points — Arterial closure device used: Femoseal® (Terumo)
  Arms: Arterial closure device used is Femoseal® (Terumo)

SUMMARY:
Over the past years, arterial closure systems have tended to replace manual compression to ensure hemostasis at femoral artery puncture points. Arterial closure systems reduce hemostasis and patient immobilization times, thus enabling early resumption of walking. These devices have contributed extensively to the development of outpatient stays for cardiology, vascular and neuro-radiology procedures.

However, main arterial closure devices use different technology to close the arterial puncture point. For some, hemostasis is achieved by sealing the arteriotomy between two discs (an inner and an outer). For others, they are designed to close puncture sites delivering a single monofilament polypropylene suture mediated by needles.

The investigators hypothesis is based on a different efficacy between both arterial closure devices for peripheral arterial disease (PAD) patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Patient with peripheral arterial disease
* Endovascular examination or treatment compatible with a 5F to 7F sheath
* Walking ability
* Patient affiliated with a social security scheme
* Patient's signed informed consent form

Exclusion Criteria:

* Under-age patient
* Patient of age, but under legal guardianship or care
* Contraindication to endovascular treatment
* Use of a 8F or greater sheath
* Morbidity contraindicating same-day walking
* History of ipsilateral open common femoral artery surgery
* Stent at the puncture site
* Radial or brachial puncture
* Antegrade femoral puncture
* Acute ischemia
* Life expectancy of less than one month
* Patient refusal to take part in the study
* Participation in another therapeutic trial
* Pregnant woman
* Allergy to clopidogrel or aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Technical success defined as hemostasis at the puncture site without major complications. | Hour 5

SECONDARY OUTCOMES:
Occurrence of major cardio-vascular events | Month 1
Occurrence of major punctured femoral artery events during the perioperative period | Hour 5
Occurrence of minor punctured femoral artery events during the perioperative period | Hour 5
Walking ability | Hour 5
  Time before restart of the ambulation measured in minutes from when the sheath of the introducer of the arterial closure system is removed and the moment when the patient is able to walk 100 meters without the recurrence of bleeding.
Quality of life evaluation (EQ-5D) | Month 1
Cost-Outcome Ratio of patient care with FemoSeal® (St Jude) and Proglide® (Abbott) | Month 1
  The measure of effectiveness will be the utility obtained from the EQ-5D quality of life questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHAILLOU, Doctor, Study Chair — Nantes University Hospital
Locations (6):
- France (6):
  - CHU Angers, Angers
  - CHU Brest, Brest
  - CH de Cholet, Cholet
  - CHD La Roche-sur-Yon, La Roche-sur-Yon
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goueffic Y, Picquet J, Schneider F, Kaladji A, Marret O, Muller L, Guyomarc'h B, Riche VP, Chaillou P, Guillou M, Nasr B. A Randomized Trial Comparing Polymer Versus Suture-Based Vascular Closure Devices for Arterial Closure Following Lower-Limb Arterial Endovascular Revascularization. Cardiovasc Intervent Radiol. 2021 Dec;44(12):1883-1892. doi: 10.1007/s00270-021-02940-z. Epub 2021 Aug 13. PMID 34386892